CLINICAL TRIAL: NCT05435911
Title: Comparison of Recovery From General Anesthesia in Remimazolam With Flumazenil Compared to Propofol-based Total Intravenous Anesthesia in Patients Undergoing Breast Cancer Surgery: a Randomized Controlled Trial
Brief Title: Comparison of Recovery From General Anesthesia in Remimazolam With Flumazenil vs. Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Remimazolam_recovery
Record Dates: First submitted 2022-06-07; First posted 2022-06-28 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Recovery
Keywords: recovery; remimazolam; flumazenil; propofol; safety
MeSH Terms: interventions — Injections, Intravenous; Powders; Flumazenil; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam with flumazenil (Experimental): Patients allocated to remimazolam with flumazenil group receive remimazolam as the main anesthetics during general anesthesia and then flumazenil administration at the end of anesthesia. Remifentanil continuous infusion can be used for hemodynamic stability and analgesia.
  Interventions: Drug: REMIMAZOLAM BESYLATE 2.5 Mg in 1 mL INTRAVENOUS INJECTION, POWDER, LYOPHILIZED, for SOLUTION [BYFAVO]; Drug: Flumazenil
- Propofol-based total intravenous anesthesia (Active Comparator): Patients allocated to the propofol-based total intravenous anesthesia group receive propofol as the main anesthetics during general anesthesia until the end of anesthesia. Remifentanil continuous infusion can be used for hemodynamic stability and analgesia.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: REMIMAZOLAM BESYLATE 2.5 Mg in 1 mL INTRAVENOUS INJECTION, POWDER, LYOPHILIZED, for SOLUTION [BYFAVO] — Remimazolam Besylate is used as an intervention drug for general anesthesia, followed by flumazenil administration at the end of anesthesia, compared to propofol-based total intravenous anesthesia during breast cancer surgery under general anesthesia
  Other Names: Remimazolam Besylate
  Arms: Remimazolam with flumazenil
Drug: Flumazenil — Flumazenil is used as an additional intervention drug to facilitate emergence from general anesthesia in the Remimazolam with Flumazenil group.
  Arms: Remimazolam with flumazenil
Drug: Propofol — Propofol is used as an active comparator drug for general anesthesia until the end of anesthesia, to be compared to remimazolam besylate during breast cancer surgery under general anesthesia.
  Arms: Propofol-based total intravenous anesthesia

SUMMARY:
This prospective randomized trial aims to compare recovery time from discontinuation of remimazolam followed by flumazenil administration vs. propofol-based total intravenous anesthesia in patients undergoing breast cancer surgery.

DETAILED DESCRIPTION:
Adult patients undergoing breast cancer surgery are randomized to receive either remimazolam with flumazenil or propofol-based total intravenous anesthesia. When the surgery is ended, anesthetic agents are discontinued. The study's primary outcome is a comparison of the time to the first eye-opening response to the doctor's command from the discontinuation of anesthetic agents between the groups. Secondary outcomes include the time from anesthetics off to extubation/discharge from operating room (OR), BIS score at eye-opening/extubation/discharge from OR, the incidence of emergence agitation at OR, the PAT score, the modified Aldrete score, modified OAA/S (Observers Assessment of Alertness/Sedation Scale) after PACU administration. In addition, the investigators investigate postoperative pain score at 10/20/30 minutes and postoperative nausea and vomiting after PACU administration, Korean version of quality of recovery-15 in postoperative 24 hours, postoperative pain score and postoperative nausea and vomiting, postoperative opioid consumption in postoperative 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, age >19, scheduled for breast cancer surgery under general anesthesia

Exclusion Criteria:

* Patients who are not alert before procedure
* Day surgery
* BMI ≥35
* Hemodynamicaly unstable patients before procedure
* Patients with history of neromuscular disease or drug use affecting neuromuscular function.
* Patients with history of adverse reaction of allergic reaction to study drugs
* Patients who are anticipated to be unable to remove supraglottic airway or endotracheal tube due to severe dyspnea or need for mechanical ventilatory support
* Use of sedatives (anxiolytics, psychoactive medication, antidepressants, hypnotics) within 24 h
* Known galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Alcohol or drug dependence
* Organic brain disorder
* Patients with hypersensitive to beans or peanut
* Patients who refuse to participate

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Time to eye opening (minute) | 20 minutes after anesthesia emergence
  The time to the first eye-opening response to the doctor's command from the discontinuation of anesthetic agents

SECONDARY OUTCOMES:
Time to emergence (minutes) | 20 minutes after anesthesia emergence
  The time from anesthetics off to extubation/discharge from operating room
Bispectral index score (Score) | During 20 minutes after anesthesia emergence (3 point : Time from anesthetics off to eye opening/extubation/discharge from operating room)
  A BIS score quantifies changes in the electrophysiologic state of the brain during anesthesia. In patients who are awake, a typical BIS score is 90 to 100. Complete suppression of cortical activity results in a BIS score of 0, known as a flat line. Lower numbers indicate a higher hypnotic effect.
Incidence of emergence agitation at operating room (n(%)) | Time Frame: 20 minutes after anesthesia emergence
  Ricker sedation agitated scale ≥5 was defined as emergence agitation, (1-7)
The modified Aldrete score (Score) | 30 minutes after post anaestheisa care unit adminstration
  The modified Aldrete score (0-10), Score ≥9 was defined as the possibility of discharge from PACU
The modified Observers Assessment of Alertness/Sedation Scale (Score) | 30 minutes after post anaestheisa care unit adminstration
  The modified Observers Assessment of Alertness/Sedation Scale (0-5), Score 5 was defined as respond readily to name spoken in normal tone.
Postoperative Pain (score) | 10/20/30 minutes after post anaestheisa care unit administation
  Numerical rating scales score (0-10) of pain, The higher score was defined as severe pain
Postoperative opioid consumption (The number of analgesic use) | from post anaestheisa care unit administation to post anaestheisa care unit discharge (during 30-40 minutes, upto 1 hours)
  Postoperative opioid requirement
Postoperative nausea and vomiting (The incidence of PONV, n(%)) | from post anaestheisa care unit administation to post anaestheisa care unit discharge (during 30-40 minutes, upto 1 hours)
  Postoperative nausea and vomiting
Postoperative quality of recovery (score) | upto 24 hours
  Korean version of quality of recovery-15, The higher score was defined as good satisfaction.
Postoperative opioid consumption (The number of analgesic use) | upto 24 hours
  Postoperative opioid requirement
Postoperative Pain (score) | upto 24 hours
  Numerical rating scales score (0-10) of pain, The higher score was defined as severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee J, Kim DH, Ju JW, Nam K, Cho YJ, Jeon Y, Lee S. Comparison of recovery profiles between total intravenous anaesthesia with propofol or remimazolam reversed with flumazenil in patients undergoing breast surgery: A randomised controlled trial. Eur J Anaesthesiol. 2024 Mar 1;41(3):199-207. doi: 10.1097/EJA.0000000000001951. Epub 2024 Jan 11. PMID 38205822